CLINICAL TRIAL: NCT00227292
Title: Cipralex in Treatment of Depressive Symptoms and Chronic Back Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Mutual agreement between Sponsor and Investigator.
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Dr. Preuss, Prof., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT Nr.2005-001673-10; JOS 05/01 (Other: Eudra); NCT00294333 (obsolete NCT alias)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Low Back Pain; Depression
Keywords: Low back pain; Depression
MeSH Terms: conditions — Low Back Pain; Depression | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 2, II (Placebo Comparator): Placebo 10mg per day for the first week, then 20mg per day till the end of study.
  Interventions: Drug: Placebo
- A, 1 (Experimental): Escitalopram 10mg per day for the first week, then 20mg per day till the end of study.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10mg per day for the first week, then 20mg per day till the end of study.
  Other Names: Cipralex
  Arms: A, 1
Drug: Placebo — Placebo 10mg per day for the first week, then 20mg per day till the end of study.
  Arms: A, 2, II

SUMMARY:
Chronic low back pain (CLBP) is one of the most frequent forms of chronic pain and can result in significant functional impairment. This is often associated with major depression too. Previous research reported significant beneficial effects of antidepressant medication in alleviating depression and pain intensity. The aim of this study is to evaluate the efficacy of Escitalopram, a new kind of Selective Serotonin Reuptake Inhibitor (SSRI) in patients with CLBP in a prospective, randomized and double-blind clinical trial. The main hypothesis is:

-in comparison to placebo, subjects with CLBP and Cipralex report a significant reduction in depressive symptoms (>= 50% of HAMD questionnaire) after 4 weeks of treatment.

DETAILED DESCRIPTION:
Pain is an unpleasant sensory and emotional experience. Chronic pain, including chronic low back pain, represents a major public health problem. Risk factors of chronicity of low back pain include high levels of psychological distress prior to or during the episode, premorbid association with work status or employment dissatisfaction, unemployment, poor self-rated health and low levels of physical activity. Other psychosocial features are poor social and educational status, previous sexual or physical abuse. Furthermore, mechanical strain on the spine from heavy lifting, repetitive lifting, twisting and vibration, including driving increase the risk. Static work postures, prolonged standing or walking, road traffic accidents and falls are also significantly related.While there is little evidence for a specific personality profile, stress, distress, anxiety, mood disorders and depression were consistently related to neck and back pain.

CLBP is associated with significant disability, functional impairment, high rates of psychiatric symptoms including anxiety and depression, and loss of other physical roles. These may produce social and functional problems, which include reduced earning capacity, unemployment and family disharmony. Chronic pain is also associated with loss of self confidence and self-esteem, leading to social withdrawal and social isolation. Men with CLBP have significantly higher lifetime rates of major depression, alcohol use disorder and major anxiety disorder. After age of pain onset, CLBP subjects had over 9 times the risk of developing major depression.

Depression is believed to be mediated by 5-HT and norepinephrine through the raphe nucleus and locus coeruleus projections to the cerebral cortex and forebrain limbic systems, whereas pain is believed to be mediated in part through descending 5-HT and norepinephrine pain pathways that provide inhibitory input to the dorsal horn neurons in the spinal cord. Global deficiences in 5-HT or norepinephrine neurotransmission would be predicted to affect both mood and pain thresholds, possibly accounting for the hgh comorbidity of painful symptoms in patients with depression.Accordingly, enhancement of both neurotransmitter or 5-HT alone would be expected both to improve symptoms of depression and to normalize pain thresholds.

In antidepressant treatment of CLBP, only 2 studies were published using SSRIs. One reported significantly higher pain intensity reduction in maprotilin group compared to paroxetine and placebo. The other showed no effect of paroxetine on depression or pain. Patients on SSRI, however, reduced the amount of analgesic medication.

ELIGIBILITY:
Inclusion Criteria:

* In- and out-patients at KH Bethanien, Greifswald, presenting with non-specific chronic low back pain lasting longer than 6 months (assessed with VAS and OLBPQ rev.)
* Age from 18 to 65 years
* Depressive symptoms (HAMD scores >10)
* Significant disability in daily living tasks (Owestry Disability Index >30%)
* Medication with nonsteroidal anti-inflammatory drugs.

Exclusion Criteria:

* Other significant Axis I disorders, including psychosis, eating disorders, substance use disorders or recent suicidal behavior.
* Systemic inflammatory disorder, malignancy, other acute medical or neurological disorders, recent surgery within 12 months.
* Medication with opioids, corticosteroids, other psychotropic medication except Temazepam.
* History of gastric ulcer, gastritis or gastric bleeding.
* Known allergy or intolerance to Citalopram or Cipralex.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
In comparison to placebo-treated patients, patients with treated with Cipralex report a significant reduction in depressive symptoms (>= 50% HAMD score) after 4 weeks of treatment. | 4 weeks

SECONDARY OUTCOMES:
In comparison to placebo, subjects treated with Cipralex report a significant reduction in pain intensity (>= 50% reduction of pain questionnaire score or VAS) after 12 weeks of treatment. | 12 weeks
In comparison with placebo, subjects treated with Cipralex report a significant improvement in physical and everyday functioning after 12 weeks of treatment. | 12 weeks
Personality traits do not have a significant influence on outcome regarding depressive traits, pain intensity and functioning. | 12 weeks
Personality disorders are significantly influencing worse outcome regarding depressive traits, pain intensity and functioning. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich W Preuss, MD, Principal Investigator — Krankenhaus Bethanien gGmbH
Locations (1):
- Martin-Luther-University Halle, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Result] Dickens C, Jayson M, Sutton C, Creed F. The relationship between pain and depression in a trial using paroxetine in sufferers of chronic low back pain. Psychosomatics. 2000 Nov-Dec;41(6):490-9. doi: 10.1176/appi.psy.41.6.490. PMID 11110112
- [Result] Atkinson JH, Slater MA, Wahlgren DR, Williams RA, Zisook S, Pruitt SD, Epping-Jordan JE, Patterson TL, Grant I, Abramson I, Garfin SR. Effects of noradrenergic and serotonergic antidepressants on chronic low back pain intensity. Pain. 1999 Nov;83(2):137-45. doi: 10.1016/s0304-3959(99)00082-2. PMID 10534584